CLINICAL TRIAL: NCT03787121
Title: Estimation of Economic Consequences Linked With Different Care Management Pathways of Differentiated Thyroid Cancers : Involvement of Overtreatment
Brief Title: Estimation of Economic Consequences Linked With Different Care Management Pathways of Differentiated Thyroid Cancers
Acronym: ECO-THYR
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/17/0378
Record Dates: First submitted 2018-12-24; First posted 2018-12-26 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Thyroid Cancer
Keywords: health economics; care management pathways; overtreatment
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: care management pathways — different care management pathways, including thyroidectomy, iode 131, hormonal treatment and type of follow up

SUMMARY:
The incidence of Thyroid Cancer (TC) has increased over the last thirty years, in France and worldwide. This increase is mainly due to good prognosis microPapillary TC (mPTC). Sixty percent of diagnosed cancers are considered as over-diagnosed, leading to an over-treatment of these cases. The increase of diagnosis of mPTC and its treatment inevitably leads to an increase of medical resources consumption and corresponding costs.

The primary aim of this study is to estimate the cost related to different care management pathway of TC patient during a lifetime period using a multi-state Markov model.

This is a retrospective, observational population based cohort study, using data from a cohort study of TC patients implemented by the ONCOMIP network which initially aimed to perform an audit of clinical practices for the management of TC, and from database of the French social health insurance of Midi-Pyrenees region to calculate observed costs of TC management during 24 months.

ELIGIBILITY:
Inclusion Criteria:

* all patients with a good prognosis of the TC
* diagnosed in 2014
* whose medical file discussed in MultiDisciplinary Team Meeting (MDTM) in Midi-Pyrenees

Exclusion Criteria:

* patients whose surgical management was carried out outside Midi Pyrenees are excluded and other morphological types are excluded (medullar, anaplastic, lymphomas, sarcomas)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Evathyr database collected by the Oncomip network: Cohort describing the initial management of 423 patients with TC diagnosed in 2014 and passed in the process of Multidisciplinary Team Meeting (MTM).
Sampling Method: Non-Probability Sample
Enrollment: 361 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
cost related to the different management pathways of TC patient | 24 months
  estimate the cost related to the different management pathways of TC patient during a lifetime period using a multi-state Markov model

CONTACTS AND LOCATIONS:
Overall Officials: Nadège Costa, PhD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University HospitalToulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No